CLINICAL TRIAL: NCT03826420
Title: Swift, Certain, and Fair: Reducing Recidivism and Improving Outcomes for Alcohol and Drug Users on State Parole
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Botec Analysis, LLC (Industry)
Collaborators: Pennsylvania Department of Corrections (Unknown); Bureau of Justice Assistance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BOTEC PADOC SCF
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Substance Abuse; Criminal Behavior
MeSH Terms: conditions — Substance-Related Disorders; Criminal Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants (parolees) will not be notified as to which arm they are enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Secure Confinement Group (Experimental): Parolees assigned to this group will be assigned sanctions that include secure confinement.
  Interventions: Behavioral: SCF Supervision with Secure Confinement Sanctioning
- Work Release Group (Experimental): Parolees assigned to this group will be assigned sanctions that include work-release.
  Interventions: Behavioral: SCF Supervision with Work Release Sanctioning
- GPS Supervision Group (Experimental): Parolees assigned to this group will be assigned sanctions that include GPS supervision.
  Interventions: Behavioral: SCF Supervision with GPS Supervision Sanctioning
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: SCF Supervision with Secure Confinement Sanctioning — Parolees assigned to this group will, in the face of a violation, be given a sanction that involves secure confinement.
  Arms: Secure Confinement Group
Behavioral: SCF Supervision with Work Release Sanctioning — Parolees assigned to this group will, in the face of a violation, be given a sanction that involves work-release.
  Arms: Work Release Group
Behavioral: SCF Supervision with GPS Supervision Sanctioning — Parolees assigned to this group will, in the face of a violation, be given a sanction that involves GPS supervision.
  Arms: GPS Supervision Group

SUMMARY:
This research project will study the outcomes of medium- to high-risk parolees with a history of substance abuse in Alleghany County, Pennsylvania supervised under Swift-Certain-Fair parole.

The research goals are to:

* Determine the effectiveness of SCF parole in reducing recidivism among medium- to high-risk parolees with a history of substance abuse in Pennsylvania.
* Determine the minimum effective sanction in response to a violation that will bring parolees into compliance with the conditions of their parole.

ELIGIBILITY:
Inclusion Criteria:

* Assigned to the Pittsburgh District
* Allegheny County resident
* Has at least 2 years left on supervision
* Had a prior drug or alcohol related sanction

Exclusion Criteria:

* Sex offender
* Reentrants assigned to the Special Needs Unit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Revocation Rate | 9 Months
  Percentage of subjects in each condition who are revoked from parole and returned to prison

SECONDARY OUTCOMES:
Days Incarcerated | 9 Months
  Total number of days incarcerated in jail or prison per parolee
New Charges | 9 Months
  Number of new charges per parolee
Percent Positive Drug Tests | 9 Months
  Percentage of random and scheduled drug tests that result in a positive reading for illicit drugs

CONTACTS AND LOCATIONS:
Overall Officials: Mark AR Kleiman, Principal Investigator — BOTEC Analysis

IPD SHARING:
Plan to Share IPD: Undecided